CLINICAL TRIAL: NCT01869101
Title: A Multicenter, 26-Week, Prospective Observational Study in Adult Patients With Prediabetes Assessing Patient Treatment and Outcomes in Community-Based Clinical Practice
Brief Title: Prospective Observational Study Assessing Treatment and Outcomes of Patients With Prediabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tethys Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TET2013-001
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Prediabetes
Keywords: Prediabetes; Diabetes prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to assess the treatment and outcomes of patients with prediabetes in community-based clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of prediabetes based on hemoglobin A1C and/or fasting plasma glucose
* Established patient of Principal Investigator's clinical practice
* BMI greater than or equal to 25 kg/m2
* Physically able to participate in a diabetes prevention program

Exclusion Criteria:

* Has prior diagnosis of diabetes
* Is pregnant or is planning to become pregnant in the next 6 months
* Is currently taking a medication prescribed for diabetes prevention
* Is currently enrolled in a formal diabetes prevention or weight loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: U.S.-based primary care practices
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Diabetes prevention treatment decisions by physician | 6 months
  The physician's clinical decision (e.g., counseling, referral to dietician, diet and exercise program) at the time of study subject visits will be recorded, summarized descriptively, and ranked in order of intensity based on pre-specified criteria.

SECONDARY OUTCOMES:
Subject initiation and persistence with diabetes prevention interventions | 6 months
  Whether or not the study subject initiates physician recommended diabetes prevention efforts and study subjects persistence with prevention recommendations will be assessed throughout the 6-month duration of the study.

OTHER OUTCOMES:
fasting glucose | 6 months
Hemoglobin A1C | 6 months
Blood pressure | 6 months
Body weight | 6 months
BMI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Frias, M.D., Study Director — Tethys Bioscience; David G Marrero, Ph.D., Study Chair — Indiana University School of Medicine